CLINICAL TRIAL: NCT07247435
Title: Role of Computed Tomography in Diagnosis of Syndromic and Non Syndromic Tetralogy of Fallot
Brief Title: Role of CT in Tetralogy of Fallot Diagnosis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Benyamin Adel Abdullah Gaballah, RD, Assiut University
Other Study IDs: Cardiac CT
Record Dates: First submitted 2025-09-24; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cardiac CT TOF
MeSH Terms: interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Computed tomography — Radiological device

SUMMARY:
To evaluate the role of MSCT in diagnosis and surgical planning in tetralogy of Fallot cases.

DETAILED DESCRIPTION:
Role of Computed tomography (CT) : CT has become an indispensable imaging modality in the comprehensive evaluation and management of Tetralogy of Fallot (ToF). While echocardiography remains the initial diagnostic tool, CT offers unparalleled spatial resolution and the ability to generate high-quality, three-dimensional reconstructions of both intracardiac and extracardiac anatomy. This is particularly valuable for identifying associated anomalies such as major aortopulmonary collateral arteries (MAPCAs), anomalous coronary artery origins, and variations in pulmonary artery branching patterns that can significantly influence surgical decision-making. Preoperatively, CT enables precise assessment of the severity and extent of right ventricular outflow tract obstruction, ventricular septal defect morphology, and the relationship of the overriding aorta to the interventricular septum.

Overall, CT complements other imaging modalities by providing a fast, accurate, and comprehensive anatomical roadmap that guides surgical planning, informs long-term follow-up, and aids in the early detection of complications. Its role is particularly pronounced in complex and syndromic cases of ToF, where anatomical variations are more common and precise preoperative mapping is critical for successful outcomes.

ELIGIBILITY:
Inclusion Criteria:

- patients aged 1 day up to 12 years Confirmed diagnosis of tetralogy of Fallot. Patients with tetralogy of Fallot as apart from genetic syndrome.

Exclusion Criteria:

* Patients with other isolated congenital heart anomalies Previously operated cases of tetralogy of Fallot.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with tetralogy of Fallot either syndromic or non syndromic
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2028-09-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Anatomical anomalies identification | 3 years
  Identification cardiac and extra-cardiac anatomical anomalies

CONTACTS AND LOCATIONS:
Overall Officials: WAGEEH Abd el-hafeez, Principal Investigator — Assiut University

REFERENCES:
- [Background] Hoffman JI, Kaplan S. The incidence of congenital heart disease. J Am Coll Cardiol. 2002 Jun 19;39(12):1890-900. doi: 10.1016/s0735-1097(02)01886-7. PMID 12084585
- [Background] Freeman SB, Bean LH, Allen EG, Tinker SW, Locke AE, Druschel C, Hobbs CA, Romitti PA, Royle MH, Torfs CP, Dooley KJ, Sherman SL. Ethnicity, sex, and the incidence of congenital heart defects: a report from the National Down Syndrome Project. Genet Med. 2008 Mar;10(3):173-80. doi: 10.1097/GIM.0b013e3181634867. PMID 18344706